CLINICAL TRIAL: NCT06151353
Title: Investigation of the Performance of Radiofrequency Echographic Multispectrometry (REMS) to Assess Bone Density and Bone Fragility in People Living in England, Scotland and Wales
Brief Title: Performance of REMS Bone Densitometry in a British Population
Status: Enrolling by invitation | Type: Observational
Sponsor: OsteoscanUK Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: REMS001
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Bone Densitometry
Keywords: REMS; Bone densitometry; Bone mineral density; Bone fragility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: REMS — Bone health assessment using REMS, an ultrasound technology developed to measure bone mineral density and bone toughness without ionising radiation

SUMMARY:
Radiofrequency echographic multispectrometry (REMS) is a recently developed technology that uses ultrasound to assess bone density and bone quality. It was launched in 2018 since when OsteoscanUK Ltd has offered a clinical bone health service using a REMS scanner. REMS is an alternative to x-ray based dual energy x-ray absorptiometry (DEXA) scans which are considered the "Gold Standard" for clinical densitometry. REMS is unique in offering not only bone density but also bone quality assessments in real time for both the spine and hip.

DETAILED DESCRIPTION:
All patients who undergo REMS scans through the OsteoscanUK bone health service, are provided with a comprehensive consent form at least two weeks ahead of the scan and are required to complete the form before the scan is performed. The process allows consent for use of their anonymized data for research purposes and is consistent with the General Data Protection Regulations in the United Kingdom (UK) and Europe.

Once a REMS scan has been completed, data is extracted from the report and is entered into an Microsoft Excel spreadsheet. Data collected includes: age, age at menopause if female, current Fracture Risk Assessment (FRAX) score, body mass index, bone mineral density results for the hip and spine, fragility scores for the hip and spine and any history of a fragility fracture.

The spreadsheet is securely stored on a password protected server and the data controller is the only person with access. Associate researchers will be provided with data from exports of parts of the spreadsheet to allow them to carry out statistical analyses. All such data will be managed on secure computers controlled by OsteoscanUK.

Results of the data analysis will be collected, analysed and presented as a series of papers to be published in peer review journals. At the time of submission of such papers, the anonymized data set would be made available to the journal editors and reviewers as required for the purposes of publishing.

ELIGIBILITY:
Inclusion Criteria:

* All women over the age of 20 years presenting for a REMS scan

Exclusion Criteria:

* Lack of consent for the procedure and for the anonymised data to be stored and used for research; Previous bilateral total hip replacements; un controlled spasticity following a neurological injury of development of a neurodegenerative condition

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — All females undergoing REMS scans
Study Population: Female patients in Great Britain over the age of 20 years who have clinical indications for a REMS bone health assessment.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2030-11-20 (Estimated); Study Completion 2031-05-20 (Estimated)

PRIMARY OUTCOMES:
Longitudinal assessment of the change in bone mineral density (BMD) and bone toughness (Fragility Score) and correlation with fragility fracture status, age, menopausal status and body mass index, | 5 years for collection of sufficient data for meaningful analysis
  Analysis of the change in bone health parameters measured by REMS from the start of the study until final follow-up which will be at least 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nick Birch, FRCS (Orth), Principal Investigator — Director of OsteoscanUK
Locations (1):
- Bragborough Hall Health Centre, Daventry, Northamptonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided